CLINICAL TRIAL: NCT05098691
Title: Serum Nectin-4 Levels in Patients With Early Onset Preeclampsia
Brief Title: Early Onset Preeclampsia and Nectin-4
Status: Completed | Type: Observational
Sponsor: Hatice Akkaya (Other Government)
Responsible Party: Sponsor-Investigator, Hatice Akkaya, associate professor, Kayseri Education and Research Hospital
Organization: Kayseri Education and Research Hospital (Other Government)
Other Study IDs: KAEK/2020.05.13
Record Dates: First submitted 2021-10-16; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Pre-Eclampsia; Early Onset Preeclampsia; Oxidative Stress; Immunologic Diseases in Pregnancy
Keywords: early onset preeclampsia; nectin-4; advers pregnancy outcome; hypertansion
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Early onset Preeclampsia ): 43 cases The groups were matched for gestational age and gravidity.
  Interventions: Diagnostic Test: serum marker levels
- Group 2 ( Healthy pregnant woman) control group: 41 cases The groups were matched for gestational age and gravidity
  Interventions: Diagnostic Test: serum marker levels

INTERVENTIONS:
Diagnostic Test: serum marker levels — two groups comparisons

SUMMARY:
Early-onset Preeclampsia (PE) is a pregnancy disorder which may present with adverse pregnancy outcomes. Nectin-4 is an adhesion molecule mainly expressed in placenta. This study aimed to evaluate the relationship between early onset Preeclampsia and serum Nectin 4 levels.

DETAILED DESCRIPTION:
Preeclampsia is assumed as a two-stage disorder arising from defective trophoblast invasion and failure of spiral artery remodeling as the main step responsible for the pathogenesis. PE is classified according to the disease onset time as early-onset PE before 34 weeks and late-onset PE after 34 weeks. Late-onset PE is more commonly seen and accepted as a mild maternal reaction to pregnancy. In early-onset PE, unlike the late-onset, due to the improper placental invasion, the diffuse placental ischemia and the resulting oxidative stress begin at early gestation. Thus, the early-onset PE may result in severe disease leading to perinatal and maternal morbidity and mortality.

The nectins are calcium-independent immunoglobulin-like celladhesion molecules and have a pivotal role at cellular junctions, as well as physiological regulations(8). Placenta expressesfor types of nectins; nectin-1, nectin-2, nectin-3, and nectin-4. They are localized at tight junctions and gap junctions of syncitiotrophoblasts(9). Nectin-4 is a relatively novel member of nectin family which has been detected only in placenta and airway epithelium in healthy subjects.

Despite, there has been no study published yet to reveal the soluble nectin-4 levels in preeclampsia as well as in early onset disease. In this study, we aimed to investigate the serum nectin-4 levels in early-onset preeclampsia in comparison of the healthy pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* spontaneous,
* singleton pregnancies
* above the 24 weeks of gestations
* positive fetal cardiac activity

Exclusion Criteria:

* multiple gestations,
* chronic hypertension
* hypothyroidism
* known malignancy,- diabetes mellitus,
* presence of fetal or maternal infection,
* clinical signs of chorioamnionitis (maternal fever, vaginal discharge, fetal tachycardia),
* hepatic or renal failure
* Placenta previa or pregnancies accompanied congenital fetal abnormalities or aneuploidies

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Comparison to the level of soluble nectin-4 in early-onset PE, compared to healthy pregnancies
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
serum nectin-4 levels | 1 hour
  ng/ml

SECONDARY OUTCOMES:
BMI (body mass index) | 5 minute
  kg/m2
Tansion Arterial | 5 minute
  mm Hg

CONTACTS AND LOCATIONS:
Locations (1):
- Hatice Akkaya, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
If needed
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: journals editors request